CLINICAL TRIAL: NCT04117802
Title: Impact of Free Sugar Replacement by Maple Syrup on Prevention of Metabolic Disorders Associated With Overweight in Humans : Role of Gut Microbiota
Brief Title: Effects of Maple Syrup on Gut Microbiota Diversity and Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, André Marette, Professor, Laval University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ERABLE-21793
Record Dates: First submitted 2019-09-30; First posted 2019-10-07 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Overweight; Microbiota; Endotoxemia; Metabolic Syndrome; Non-Alcoholic Fatty Liver Disease; Insulin Resistance
MeSH Terms: conditions — Overweight; Endotoxemia; Metabolic Syndrome; Non-alcoholic Fatty Liver Disease; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maple (Experimental)
  Interventions: Other: Maple syrup
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Maple syrup — Substitution of refined sugar by an equivalent quantity of maple syrup (5% of daily energy intake) in the participant diet. A dietitian will help study subjects to target added sugar sources in their usual diet and suggest ways to substitute it with maple syrup.
  Arms: Maple
Other: Placebo — Substitution of refined sugar by an equivalent quantity of maple-flavored sucrose syrup (5% of daily energy intake) in the participant diet. A dietitian will help study subjects to target added sugar sources in their usual diet and suggest ways to substitute it with the placebo (sucrose syrup).
  Arms: Placebo

SUMMARY:
It has been suggested that the actual obesity epidemy is related to chronic overconsumption of added or free sugars. The increasing popularity of artificial sweeteners attest the population willingness to reduce added sugars intake and to use alternatives to alleviate health impact of free sugar overconsumption. However, recent findings suggest that artificial sweeteners may rather contribute to obesity epidemy and its associated adverse health effects, potentially via a negative impact on gut microbiota. It has been shown in various studies that, for the same amount of sucrose, unrefined sugars (such as maple syrup) are associated with favorable metabolic effects. The polyphenols contained in maple syrup, especially lignans, could contribute to these positive effects. Indeed, the strong impact of those biomolecules on the modulation of gut microbiota and on gastro-intestinal and metabolic health has been demonstrated in several studies. It is therefore highly relevant to test the hypothesis that the substitution of refined sugar by an equivalent amount of maple syrup (5% of daily energy intake) result in a lesser metabolic deterioration, by the modulation of maple syrup on gut microbiota, than the one observed with refined sugar.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 23 and 40 kg/m2
* At least one of the following: Fasting triglyceride > 1,35 mmol/L, Fasting insulinemia > 42 pmol/L, fasting glycemia between 5,5 and 6,9 mmol/L and glycated haemoglobin (HbA1c) between 5.7 and 6.4 %
* Understanding of spoken and written french
* Accept to follow study instructions
* If there is natural health product consumption, the dose and frequency of consumption must be stable since 3 months or more

Exclusion Criteria:

* Smoking
* Any metabolic disorder requiring medication or affecting glucose or lipid metabolism
* Aversion for maple taste
* Allergy or intolerance for maple syrup or for an ingredient of the placebo syrup
* Alcohol consumption of > 2 drinks / day
* Weight change > 5% of body weight in the last 3 months
* Being in a weight loss attempt
* Antibiotics intake in the last 3 months
* Regular probiotics intake in the last 3 months
* Major surgical operation in the last 3 months or planned in the next months
* Gastrointestinal malabsorption
* Cirrhosis
* Chronic kidney disease
* Pregnant or breastfeeding women or women planning pregnancy in the next months
* Participation in another clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Glucose homeostasis | Change between the beginning and the end of each treatment (8 weeks each)
  Evaluation of plasma glucose, insulin and c-peptide concentration using a 3-hour oral glucose tolerance test

SECONDARY OUTCOMES:
Change in Endotoxemia | Change between the beginning and the end of each treatment (8 weeks each)
  Plasma Lipopolysaccharides (LPS) and Lipopolysaccharide Binding Protein (LBP)
Change in Intestinal permeability | Change between the beginning and the end of each treatment (8 weeks each)
  Plasma zonulin
Change in Inflammation state of the tissue | Change between the beginning and the end of each treatment (8 weeks each)
  Fecal calprotectin and chromogranin
Change in Short chain fatty acids in the feces | Change between the beginning and the end of each treatment (8 weeks each)
  Measure short chain fatty acids in the feces
Change in Gut health and stool consistency | Change between the beginning and the end of each treatment (8 weeks each)
  Evaluation of gastrointestinal symptoms and stool consistency using standardized questionnaires (the gastrointestinal symptom rating scale (GSRS) and Bristol stool chart)
Change in fat accumulation in the liver | Change between the beginning and the end of each treatment (8 weeks each)
  Evaluation of fat accumulation by magnetic resonance imaging (MRI)
Change in Glucose homeostasis | Change between the beginning and the end of each treatment (8 weeks each)
  Evaluation of glycated haemoglobin
Change in Lipid profile | Change between the beginning and the end of each treatment (8 weeks each)
  Evaluation of plasma triglycerides (TG), Total cholesterol, LDL, HDL, Apolipoprotein B and free fatty acids end of two dietary treatment
Change in anthropometric measurements | Change between the beginning and the end of each treatment (8 weeks each)
  Evaluation of bmi with weight and height measurements
Change in anthropometric measurements | Change between the beginning and the end of each treatment (8 weeks each)
  Evaluation of waist circumference
Change in body composition | Change between the beginning and the end of each treatment (8 weeks each)
  Evaluation of body composition by osteodensitometry
Change in chronic inflammation | Change between the beginning and the end of each treatment (8 weeks each)
  Evaluation of plasma high sensitive C-Reactive Protein (hs-CRP)
Change in gene expression levels | Change between the beginning and the end of each treatment (8 weeks each)
  Transcriptomic analyses to investigate underlying mechanisms of action
Change in circulating levels of plasma metabolites | Change between the beginning and the end of each treatment (8 weeks each)
  Metabolomic analyses to investigate underlying mechanisms of action
Change in maple-derived metabolites present in stool | Change between the beginning and the end of each treatment (8 weeks each)
  Evaluation of metabolome: camu-camu derived metabolites, short chain fatty acids, branched chain fatty acids, bile acids, phenolic compounds
Change in blood pressure | Change between the beginning and the end of each treatment (8 weeks each)
  Evaluation of systolic and diastolic blood pressure
Change in Gut Microbiota Composition | Change between the beginning and the end of each treatment (8 weeks each)
  Gut microbiota composition will be evaluated by 16S rRNA amplicon sequencing (V3-V4 region)
Change in Gut Microbiota Composition | Change between the beginning and the end of maple syrup treatment (8 weeks)
  Gut microbiota composition will also be evaluated by whole genome sequencing
Change in Gut Microbiota alpha Diversity | Change between the beginning and the end of each treatment (8 weeks each)
  To quantify bacterial alpha diversity, Shannon's reciprocal index will be calculated
Change in Gut Microbiota alpha Diversity | Change between the beginning and the end of each treatment (8 weeks each)
  To quantify bacterial alpha diversity, Simpson's reciprocal index will be calculated
Change in Gut Microbiota beta Diversity | Change between the beginning and the end of each treatment (8 weeks each)
  Principal component analysis (PCA) will be performed on the Aitchison distance matrix to measure beta diversity.

CONTACTS AND LOCATIONS:
Locations (1):
- INAF, Université Laval, Québec, Canada

REFERENCES:
- [Derived] Morissette A, Agrinier AL, Gignac T, Ramadan L, Diop K, Marois J, Varin TV, Pilon G, Simard S, Larose E, Gagnon C, Arsenault BJ, Despres JP, Carreau AM, Vohl MC, Marette A. Substituting Refined Sugars With Maple Syrup Decreases Key Cardiometabolic Risk Factors in Individuals With Mild Metabolic Alterations: A Randomized, Double-Blind, Controlled Crossover Trial. J Nutr. 2024 Oct;154(10):2963-2975. doi: 10.1016/j.tjnut.2024.08.014. Epub 2024 Aug 18. PMID 39163971